CLINICAL TRIAL: NCT05408650
Title: Effectiveness of Aromatherapy Massage on Sleep Quality and Physiological Parameters of Post-Operative Cardiothoracic Surgery Patients
Brief Title: Effect of Aromatherapy Massage on Sleep Quality of Post-operative Cardiothoracic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Aya Ali Saad Elhusseini, Principle Investigator (Demonstrator of critical care and emergency nursing), Mansoura University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P.0237
Record Dates: First submitted 2022-05-28; First posted 2022-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Aromatherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aromatherapy massage group (Experimental): The massage will be applied to the patient's hands and feet while the patient in semi-fowler's position.
  Interventions: Other: Aromatherapy Massage
- control group (No Intervention): The patients will receive the routine care of the ICU (such as decreased movements of the staff and soft light in the area at night).

INTERVENTIONS:
Other: Aromatherapy Massage — The PI will dilute pure lavender essential oil (Lavandula angustifolia) with almond oil at a dilution rate of 2.5% and apply it to the hands and feet of the patient.
  * The massage technique including effleurage, petrissage, friction and lymphatic drainage on hands and feet will be adapted from Salvo, (2015) and Youssef and Hassan, (2017).
  * The massage will be applied to the patient's hands and feet while the patient in semi-fowler's position.
  Arms: Aromatherapy massage group

SUMMARY:
Poor sleep is common in the ICU, especially among post-operative CABG and more severely ill patients. Additionally, patients after surgery suffer from changes in physiological parameters related to ICU stressors. Pharmacological interventions for sleep improvement can both disrupt and induce sleep and have many negative side effects on intensive care patients. Therefore, this gives the green light for using complementary therapy.

DETAILED DESCRIPTION:
Critically ill patients suffer from decreased sleep quality, especially in patients who fear death and are more severely ill. The critical care experience is stressful for patients and can result in numerous physiological and psychological effects, including physiological instability as an increase in the heart rate (HR), respiration rate (RR), and risk of cardiac dysrhythmias, leading to prolonged length of stay and subsequent complications. Sleep is affected by a variety of factors, including hospitalization and the severity of the disease. Therefore, improving the sleep quality of cardiac patients is one of the most important nursing interventions.

Sleep is a circadian state characterized by the partial or total suspension of consciousness, voluntary muscle inhibition, and relative insensitivity to stimulation. Sleep quality is an individual's general satisfaction with the sleep experience, and its main components are the quantity of sleep, sleep continuity, and a reviving feeling upon awakening. Short sleep duration is defined as less than seven hours of sleep per 24-hour period.

Sleep is a biological need for many physiological processes under primary neurobiological regulation that affects many physiological systems, so sleep is necessary for the body to repair and restore itself. At least when compared to the early morning hours, an increase in parasympathetic cardiac transition during non-rapid eye movement sleep 2 makes the nighttime a period of proportional protection from cardiovascular diseases (CVD) events. Sleep and sleep disturbances affect various components of human homeostasis, including the cardiovascular system.

Cardiovascular diseases are the most common cause of death globally, taking an estimated 17.9 million lives each year. Over three-quarters of CVD deaths take place in low and middle-income countries. In the Eastern Mediterranean Region, more than 1.3 million people died of CVD, which equals one-third of all deaths annually. Sleep disturbance is a common problem in cardiac patients. Cardiac surgery patients' perceptions of their sleep in the intensive care unit (ICU) indicate that it is inadequate.

Sleep disturbance occurs in 60 to 80% of patients in the first few days after heart surgery. One of the most common causes of sleep disturbance after coronary artery bypass graft (CABG) is subsequent alterations in physiological parameters such as systolic and diastolic blood pressure (SBP and DBP), RR, and HR.

Poor sleep quality is associated with many adverse health outcomes. Accumulating evidence proposes that insufficient sleep affects basal levels of immune, inflammatory mediators, and inflammatory reactivity to stressors. In addition, there is an increase in a person's risk of health problems and the development of many chronic.

diseases. Therefore, adequate sleep is the main requirement for physical and mental health.

Physiological changes are among the most significant symptoms and signs that need to be observed in patients with cardiothoracic diseases and surgeries. ICU patients' stress and pathological conditions cause sleep disturbances, increased oxygen consumption by the heart muscles, increased sympathetic nervous system burden, tachypnea, increased HR, and neural-hormonal responses, all of which contribute to elevated blood pressure, which complicates the healing and recovery process.

Complementary and integrative therapy (CIT) has become widely known and used in nursing. It is used alongside conventional medicine. There are several non-pharmacological methods can be helpful to improve sleep in critical patients and decrease the negative factors that affect vital signs and interrupt sleep in ICUs, including reflexology, relaxation, guided imagery, aromatherapy (AT), and massage. Complementary therapies are forms of non-pharmacological methods that are cost-effective, non-invasive, and aim to increase comfort in stressful situations.

4 Aromatherapy is a biological-based therapy in CIT. It is defined as "the art and science of utilizing naturally extracted aromatic essences from plants to balance, harmonize, and promote the health of body, mind, and spirit". Accordingly, AT depends on the use of essential oils extracted from flowers and plants. Aromatherapy affects the parasympathetic nervous system, stabilizing the patient's physiological parameters and metabolism and eventually maintaining the patient's level of relaxation.

Essential oils are used in AT to reduce certain physical and psychological manifestations and provide relaxation. Additionally, scent molecules affect the limbic system of the brain, HR, BP, RR, memory, and hormones.

Massage is one of the most commonly used techniques in CIT. It is a manipulative and body-based practice type that is often given guidance by nurses and healthcare givers to patients in their daily health care. Massage promotes relaxation by physically manipulating muscles as well as physiologically by stimulating the nervous system to regulate muscle contraction . Massage is an effective method for promoting sleep quality for ICU patients.

ELIGIBILITY:
Inclusion Criteria:

Adult conscious patients ≥ 18 years of both gender

* ICU length of stay > 2 nights
* Physiologically or hemodynamically stable
* Free from skin problems and fractures in the area of massage

Exclusion Criteria:

* Patients who are on sedative drugs or narcotic analgesics
* Patients with an allergic history to lavender oil
* Mechanically ventilated patients
* History of sleep disorders
* History of mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Quality of sleep or Level of sleep as assessed by Richards-Campbell Sleep Questionnaire | 2 days
  Sleep quality will be assessed by Richards-Campbell Sleep Questionnaire which covers five aspects of sleep: depth, latency, frequency of awakening, percentage of time awake, and sleep quality.
  A total score is obtained by summing each score out of 100, then dividing the total by five and ranking the total score into three categories as follows:
  * A score from 0 mm to 33 mm indicates poor sleep
  * A score of between 33 mm to 66 mm indicates normal sleep
  * A score of over 66 mm indicates very good sleep
Physiological parameters include heart rate, respiratory rate, systolic and diastolic blood pressure, mean arterial blood pressure, and percutaneous oxygen saturation, which will be assessed by a bedside electronic monitor. | 2 days
  Physiological parameters include heart rate, respiratory rate, systolic and diastolic blood pressure, mean arterial blood pressure, and percutaneous oxygen saturation, which will be assessed by a bedside electronic monitor.